CLINICAL TRIAL: NCT01933516
Title: Phase I Trial to Assess the Safety and Pharmacokinetics of GP2013 Monotherapy Administered Weekly in Japanese Patients With CD20 Positive Low Tumor Burden Indolent B-cell Non-Hodgkin's Lymphoma
Brief Title: GP2013 in Japanese Patients With CD20 Positive Low Tumor Burden Indolent B-cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GP13-101
Record Dates: First submitted 2013-08-08; First posted 2013-09-02 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Indolent B-cell Non-Hodgkin's Lymphoma
Keywords: GP2013; Japanese; indolent B-cell non-Hodgkin's lymphoma; biosimilar; CD20; GP13-101
MeSH Terms: interventions — Rituximab

ARMS (1):
- GP2013 (Experimental)
  Interventions: Drug: GP2013

INTERVENTIONS:
Drug: GP2013 — GP2013

SUMMARY:
The purpose of this study is to evaluate safety and pharmacokinetic of GP2013 in Japanese patients with CD20 positive low tumor burden indolent B-cell NHL under weekly dosing schedule.

ELIGIBILITY:
Inclusion Criteria:

* Patient with CD20 positive low tumor burden indolent B-cell non- Hodgkin's lymphoma.
* Patient with at least one measurable lesion.
* Patient with ECOG performance status 0 or 1.

Exclusion Criteria:

* Patient who has received radiotherapy within the last 28 days prior to administration, or are not recovered from previous radiotherapy.
* Patient who has received immunotherapy, chemotherapy, antibodies and experimental treatment within the last 28 days prior to administration, or are not recovered from previous therapy.
* Patient who has mAb therapy other than rituximab as prior line of therapy.
* Patient with evidence of any uncontrolled, acute or chronic active infection (viral, bacterial or fungal).
* Patient with any other malignancy within 5 years prior to date of screening, with the exception of adequately treated in situ carcinoma of the cervix uteri, basal or squamous cell carcinoma or nonmelanomatous skin cancer.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
To evaluate safety of GP2013 | 12 weeks
  Adverse events, laboratory abnormalities
Area under the curve calculated from start of dose to the end of the dosing interval (tau) of GP2013 | 12 weeks
Maximum observed concentration of GP2013 | 12 weeks
Time to reach maximum concentration of GP2013 | 12 weeks
Minimum (trough) observed concentration during each dosing interval of GP2013 | 12 weeks
Terminal elimination rate constant calculated as the slope of the linear regression of the terminal phase of the logarithmic concentration-time profile of GP2013 | 12 weeks
Elimination half-life associated with the terminal slope of GP2013 | 12 weeks

SECONDARY OUTCOMES:
To evaluate efficacy of GP2013 | 12 weeks
  Antitumor activity
To evaluate the incidence of immunogenicity (ADA formation) against GP2013 | 12 weeks
  Immunogenicity (ADA formation)
To evaluate peripheral CD19+ B-cell count | 12 weeks
  CD19 + B-cell count

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz K.K., Study Director — Sandoz
Locations (1):
- Investigative Site, Tachikawa, Tokyo, Japan